CLINICAL TRIAL: NCT05634668
Title: Study of Sleep Disturbances and Quality of Life Among Postmenopausal Women: A Cross-sectional Study
Brief Title: Sleep and Quality of Life Among Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Rashad Youssef Soliman, Principal Investigator, Assiut University
Other Study IDs: Menopausal Sleep disturbance
Record Dates: First submitted 2022-10-27; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Sleep Disturbance; Postmenopausal Symptoms
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interviewing sheet — 1. . Interviewing sheet: It was designed by the researchers and used to obtain subjects' sociodemographic data; their age, menopausal age, gravidity, parity, BMI, residency, occupation, education level, hot flashes, sweating, and daily habits.
  2. . Menopause specific quality of life questionnaire (MENQOL): MENQOL was designed by Hilditch and used to assess the presence of menopausal symptoms, its severity, and the degree to which they adversely affect women's life. It consisted of 29 items categorized into four domains
  3. . Pittsburgh Sleep Quality Index (PSQI): The PSQI was a self-report scale consisting of 7 components and 19 questions. PSQI studies quality of sleep in the recent month.
  Other Names: Menopause specific quality of life questionnaire (MENQOL); Pittsburgh Sleep Quality Index (PSQI)

SUMMARY:
The purpose of this study is to assess the sleep quality and quality of life of the study population.

DETAILED DESCRIPTION:
Natural menopause can be defined as the cessation of menses for twelve sequential months without physiological or pathologic causes, referring to the end of a woman's reproductive capability. There is considerable variation in reporting of menopausal symptoms by women all over the world in different studies. The most common psychological symptoms was physical, mental exhaustion and Sleep disturbances. Sleep quality is affected poorly during the menopausal transition, and 40-60% of menopausal women are suffering from sleep disturbances. The causes for sleep disorders in postmenopausal women can be divided broadly into psychological and physical. However, changes in sleep patterns after menopause are frequently the result of physical factors. Sleep quality and its effect on quality of life among postmenopausal women is vital topic and the previous Literatures in this topic are deficient. So, there is a need to study sleep quality and quality of life particularly in our population where women are less aware about menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 45-70 years, married, who experienced natural menopause conﬁrmed by menstrual cessation for at least one year or a FSH level ≥40 IU/L .

Exclusion Criteria:

* women who

  1. single, widow or divorced.
  2. had an induced menopause
  3. underwent simple hysterectomy .
  4. receiving any kind of hormone therapy, antidepressants, or antipsychotics .
  5. had medical conditions such as diabetes, hypertension, cardiac disease, and thyroid disorders .
  6. had experienced any stressful events during the past year or had depressive disorders as they can mislead our results
  7. Patient refused to participate in this study.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women will be recruited from the postmenopausal population presenting to the outpatient clinics or admitted to the inpatient wards at Assiut University Hospital and their female relatives who are between 45 and 70 years of age. A woman is defined as postmenopausal if 12 months had passed after her last menstruation. Meanwhile, we will exclude women with induced menopause, who underwent a simple hysterectomy, who is currently receiving hormonal therapy, and who has medical conditions such as diabetes, hypertension, cardiac disease, and thyroid disorders, as these may mislead our results. Additionally, women who refuses to participate in this study will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The menopausal quality of life score | one hour
  scoring the menopausal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Amira Ra Youssef Soliman, Resident, Principal Investigator — Assiut University, Assiut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Minkin MJ. Menopause: Hormones, Lifestyle, and Optimizing Aging. Obstet Gynecol Clin North Am. 2019 Sep;46(3):501-514. doi: 10.1016/j.ogc.2019.04.008. Epub 2019 Jun 21. PMID 31378291
- [Background] Gozuyesil E, Gokyildiz Surucu S, Alan S. Sexual function and quality-of-life-related problems during the menopausal period. J Health Psychol. 2018 Dec;23(14):1769-1780. doi: 10.1177/1359105317742194. Epub 2017 Dec 15. PMID 29243521
- [Background] Kling JM, Kelly M, Rullo J, Kapoor E, Kuhle CL, Vegunta S, Mara KC, Faubion SS. Association between menopausal symptoms and relationship distress. Maturitas. 2019 Dec;130:1-5. doi: 10.1016/j.maturitas.2019.09.006. Epub 2019 Sep 16. PMID 31706430
- [Background] Li CC, Tsai YF, Chang TC, Chen L. Associations among menopausal symptoms, sleep and fatigue in Taiwanese women with endometrial cancer. Eur J Cancer Care (Engl). 2017 Sep;26(5). doi: 10.1111/ecc.12559. Epub 2016 Aug 21. PMID 27545107
- [Background] AlDughaither A, AlMutairy H, AlAteeq M. Menopausal symptoms and quality of life among Saudi women visiting primary care clinics in Riyadh, Saudi Arabia. Int J Womens Health. 2015 Jun 29;7:645-53. doi: 10.2147/IJWH.S84709. eCollection 2015. PMID 26170720
- [Background] Ibrahim ZM, Ghoneim HM, Madny EH, Kishk EA, Lotfy M, Bahaa A, Taha OT, Aboelroose AA, Atwa KA, Abbas AM, Mohamed ASI. The effect of menopausal symptoms on the quality of life among postmenopausal Egyptian women. Climacteric. 2020 Feb;23(1):9-16. doi: 10.1080/13697137.2019.1656185. Epub 2019 Sep 19. PMID 31533486
- [Background] Khatoon A, Husain S, Husain S, Hussain S. An Overview of Menopausal Symptoms Using the Menopause Rating Scale in a Tertiary Care Center. J Midlife Health. 2018 Jul-Sep;9(3):150-154. doi: 10.4103/jmh.JMH_31_18. PMID 30294188
- [Background] Tadayon M, Ilkhani M, Abedi P, Haghighi Zadeh M. The relationship between sleep quality and lifestyle in postmenopausal Iranian women: a cross-sectional study. Women Health. 2019 Sep;59(8):883-891. doi: 10.1080/03630242.2019.1607802. Epub 2019 Apr 28. PMID 31032743
- [Background] Baker FC, Lampio L, Saaresranta T, Polo-Kantola P. Sleep and Sleep Disorders in the Menopausal Transition. Sleep Med Clin. 2018 Sep;13(3):443-456. doi: 10.1016/j.jsmc.2018.04.011. PMID 30098758
- [Background] Weber MT, Rubin LH, Maki PM. Cognition in perimenopause: the effect of transition stage. Menopause. 2013 May;20(5):511-7. doi: 10.1097/gme.0b013e31827655e5. PMID 23615642
- [Background] Kravitz HM, Joffe H. Sleep during the perimenopause: a SWAN story. Obstet Gynecol Clin North Am. 2011 Sep;38(3):567-86. doi: 10.1016/j.ogc.2011.06.002. PMID 21961720
- [Background] Xu Q, Lang CP. Examining the relationship between subjective sleep disturbance and menopause: a systematic review and meta-analysis. Menopause. 2014 Dec;21(12):1301-18. doi: 10.1097/GME.0000000000000240. PMID 24800878
- [Background] Ali AM, Ahmed AH, Smail L. Psychological Climacteric Symptoms and Attitudes toward Menopause among Emirati Women. Int J Environ Res Public Health. 2020 Jul 13;17(14):5028. doi: 10.3390/ijerph17145028. PMID 32668726
- [Background] Kling JM, Manson JE, Naughton MJ, Temkit M, Sullivan SD, Gower EW, Hale L, Weitlauf JC, Nowakowski S, Crandall CJ. Association of sleep disturbance and sexual function in postmenopausal women. Menopause. 2017 Jun;24(6):604-612. doi: 10.1097/GME.0000000000000824. PMID 28141665
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Suleiman KH, Yates BC, Berger AM, Pozehl B, Meza J. Translating the Pittsburgh Sleep Quality Index into Arabic. West J Nurs Res. 2010 Mar;32(2):250-68. doi: 10.1177/0193945909348230. Epub 2009 Nov 14. PMID 19915205
- [Background] Moudi A, Dashtgard A, Salehiniya H, Sadat Katebi M, Reza Razmara M, Reza Jani M. The relationship between health-promoting lifestyle and sleep quality in postmenopausal women. Biomedicine (Taipei). 2018 Jun;8(2):11. doi: 10.1051/bmdcn/2018080211. Epub 2018 May 28. PMID 29806589